CLINICAL TRIAL: NCT02959502
Title: Home-Based Cognitive Remediation and Transcranial Direct Current Stimulation to Enhance Cognition in Persons With Mild Cognitive Impairment and Late Life Depression
Brief Title: Home-Based CR and tDCS to Enhance Cognition in Persons With Mild Cognitive Impairment and Late Life Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: CAMH Foundation (Other)
Responsible Party: Principal Investigator, Tarek Rajji, Chief of Geriatric Psychiatry, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 069/2016
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment; Major Depressive Disorder; Alzheimer's Dementia; Transcranial Direct Current Stimulation; tDCS
MeSH Terms: conditions — Cognitive Dysfunction; Depressive Disorder, Major; Alzheimer Disease | interventions — Transcranial Direct Current Stimulation; Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receive tDCS + CR (Experimental): Receive tDCS+CR: Over the course of 8 weeks, for 5 days a week, participants designated a 'Patient' will receive active tDCS &CR at-home. tDCS will be administered during the 2 hour CR sessions for 30 min/day. The tDCS montage will be bifrontal91 with 1 large anode placed over Fz and the cathode over Iz. The direct current will be 2 mA (current density = 0.57 A/m2). CR sessions will utilize didactic and computerized drill-based exercises which focus on practice and repetition of neurocognitive ability areas that are affected in depression such as attention, processing speed, executive function, verbal memory, and working memory. Performance feedback is given to reinforce progress and the exercises are designed to be enjoyable to complete, with titrated difficulty levels over time.
  Interventions: Other: Receive tDCS+CR
- Facilitate tDCS + CR (Experimental): Over the course of 8 weeks, for 5 days a week, participants designated a 'facilitator' will trained to deliver tDCS &CR at-home. tDCS will be administered during the 2 hour CR sessions for 30 min/day. The tDCS montage will be bifrontal91 with 1 large anode placed over Fz and the cathode over Iz. The direct current will be 2 mA (current density = 0.57 A/m2). CR sessions will utilize didactic and computerized drill-based exercises which focus on practice and repetition of neurocognitive ability areas that are affected in depression such as attention, processing speed, executive function, verbal memory, and working memory.
  Interventions: Other: Facilitate tDCS + CR

INTERVENTIONS:
Other: Receive tDCS+CR — Over the course of 8 weeks, for 5 days a week, participants designated a 'Patient' will receive active tDCS &CR at-home. tDCS will be administered during the 2 hour CR sessions for 30 min/day. The tDCS montage will be bifrontal91 with 1 large anode placed over Fz and the cathode over Iz. The direct current will be 2 mA (current density = 0.57 A/m2). CR sessions will utilize didactic and computerized drill-based exercises which focus on practice and repetition of neurocognitive ability areas that are affected in depression such as attention, processing speed, executive function, verbal memory, and working memory. Performance feedback is given to reinforce progress and the exercises are designed to be enjoyable to complete, with titrated difficulty levels over time.
  Other Names: transcranial Direct Current Stimulation (tDCS); Cognitive Remediation (CR)
  Arms: Receive tDCS + CR
Other: Facilitate tDCS + CR — Over the course of 8 weeks, for 5 days a week, participants designated a 'facilitator' will be trained to deliver tDCS &CR at-home. tDCS will be administered during the 2 hour CR sessions for 30 min/day. The tDCS montage will be bifrontal91 with 1 large anode placed over Fz and the cathode over Iz. The direct current will be 2 mA (current density = 0.57 A/m2). CR sessions will utilize didactic and computerized drill-based exercises which focus on practice and repetition of neurocognitive ability areas that are affected in depression such as attention, processing speed, executive function, verbal memory, and working memory.
  Other Names: transcranial Direct Current Stimulation (tDCS); Cognitive Remediation (CR)
  Arms: Facilitate tDCS + CR

SUMMARY:
The overall goals of this project are to assess the feasibility and impact of designing and implementing an at-home intervention aimed at preventing long-term cognitive decline and improving cognition in individuals currently at-risk for developing AD.

DETAILED DESCRIPTION:
By the time Alzheimer's Dementia (AD) and related disorders are diagnosed, the brain has sustained substantial insult that limits the efficacy of current treatments. Preventive interventions are urgently needed but the majority of prevention studies require large numbers of participants, long follow-up periods, and frequent study visits. It is not feasible for many geriatric patients to attend clinics for treatment on a daily basis due to mobility and transportation restrictions, associated costs, and lack of rural clinic locations. Interventions delivered remotely, or administered within an individual's home, allow for preventative treatments to be made accessible to a wider range of individuals. Thus, the overall goals of this project are to assess the feasibility and impact of designing and implementing an at-home intervention aimed at preventing long-term cognitive decline and improving cognition in individuals currently at-risk for developing AD. These high-risk individuals that will be targeted in this proposal are: (1) older adults with Mild Cognitive Impairment (MCI), (2) older adults with Major Depressive Disorder (MDD), and (3) older adults with MCI and MDD.

The proposed intervention combines cognitive remediation (CR) and non-invasive brain stimulation - transcranial Direct Current Stimulation (tDCS), to be delivered in the participants' home environment. Twenty couples (40 participants) will be recruited, with one member defined as the "patient" and the second member defined as the "caregiver" to the patient. These caregivers will facilitate the delivery of the study intervention (i.e., CR+tDCS). Participants with a diagnosis of MCI or MDD or both, who have a caregiver, will receive open-label, active CR+tDCS over a period of 8 weeks. Both CR and tDCS have been shown to induce neuroplasticity and improve cognition. The aim of this pilot study is to assess the feasibility of delivering these combined interventions at home.

ELIGIBILITY:
MCI Group

Inclusion:

1. Age > 60 (on day of randomization)
2. DSM-IV criteria for Mild Neurocognitive Disorder ("MCI")
3. Willingness to provide informed consent
4. MADRS score of 10 or below
5. Availability of a study partner who has regular contact with the participant
6. Ability to read and communicate in English (with corrected vision and hearing, if needed)

Exclusion:

1. Met DSM-IV criteria for Major Depressive Episode in past 10 years
2. Lifetime DSM-IV diagnosis of schizophrenia, bipolar disorder, or OCD
3. DSM-IV diagnosis of alcohol or other substances use disorder within the past 12 months
4. High risk for suicide
5. Significant neurological condition (e.g., stroke, seizure disorder, MS)
6. Unstable medical illness, (e.g., uncontrolled diabetes mellitus or hypertension)
7. Having taken a cognitive enhancer (acetylcholinesterase inhibitor or memantine) within the past 6 weeks
8. Participants taking anticonvulsants, and other psychotropic medication (see exception below) that cannot be safely tapered and discontinued. The following psychotropic medications are allowed if they have been taken at a stable dose for at least 4 weeks prior to study entry: zopiclone, trazadone, or a benzodiazepine; gabapentin, pregabalin, duloxetine, venlafaxine, or low-dose tricyclic antidepressants if prescribed for chronic pain.
9. A pace-maker or other metal implants that would preclude safe use of tDCS.

MDD Group

Inclusion:

1. Age ≥ 60 (on day of randomization)
2. Meets DSM-IV criteria for one or more MDE(s)with:

   1. an offset of 2 months to 5 years from the screening visit date. It is not necessary for this (these) episode(s) to have received medical attention

      OR
   2. an offset of 5 years or more from the screening visit date. It is necessary that at least one MDE received medical attention (e.g., previously been on one or more antidepressant(s), saw a psychiatrist, primary care physician, or had a previous hospitalization). Also, the MDE must have occurred during the participant's adult life (i.e., at 18 years of age or older).
3. MADRS score of 10 or below
4. Willingness to provide informed consent
5. Availability of a study partner who has regular contact with the participant
6. Ability to read and communicate in English (with corrected vision and hearing, if needed)

Exclusion:

1. Meets DSM-IV criteria for Major Neurocognitive Disorder ("dementia")
2. Lifetime DSM-IV diagnosis of schizophrenia, bipolar disorder, or OCD
3. DSM-IV diagnosis of alcohol or other substances use disorder within the past 12 months.
4. High risk for suicide.
5. Significant neurological condition (e.g., stroke, seizure disorder, MS)
6. Unstable medical illness (e.g., uncontrolled diabetes mellitus or hypertension)
7. Participants taking anticonvulsants, and other psychotropic medication (see exception below) that cannot be safely tapered and discontinued. In addition to any antidepressant, the following psychotropic medications are allowed if they have been taken at a stable dose for at least 4 weeks prior to study entry: zopiclone, trazodone, or a benzodiazepine; and gabapentin or pregabalin if prescribed for chronic pain.
8. Having taken a cognitive enhancer (acetylcholinesterase inhibitor or memantine) within the past 6 weeks.
9. A pace-maker or other metal implants that would preclude safe use of tDCS.

Facilitator Group

Inclusion:

1. Willingness to provide informed consent
2. Ability to read and communicate in English (with corrected vision and hearing, if needed)

   Exclusion:
3. Physical or medical illness that prevents participant from learning or administering CR + tDCS, as determined by the research team

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of training a facilitator (caregiver) to facilitate the administration of CR+tDCS to their "patient" partner as indicated by a positive response in the Perceived Competence Scale at 24 months from study baseline. | Approximately 24 months after baseline
Fidelity to delivering home-based CR+tDCS by a facilitator (caregiver) to the participant as indicated by the compliance rate during the induction phase and boosters. | Baseline and approximately 24 months after baseline
  Compliance rate is defined as the the number of sessions completed as assessed by the Session Log divided by the total number of sessions across the induction phase and boosters.

SECONDARY OUTCOMES:
Assess change in Quality of Life Scale scores among patients between baseline and at the end of the 8-week course. | Baseline and 8 weeks after baseline.
Measure the change in Quality of Life Scale scores among facilitators between baseline and at the end of the 8-week course. | Baseline to 8 weeks after baseline.
Measure the change in cognition (as indicated by a change in the Screen for Cognitive Impairment in Psychiatry) among patients between baseline and at the end of the 8-week course | Baseline to 8 weeks after baseline.
Measure the change in cognition (as indicated by a change in the Screen for Cognitive Impairment in Psychiatry) among facilitators between baseline and at the end of the 8-week course | Baseline to 8 weeks after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Rajji, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research